CLINICAL TRIAL: NCT01883934
Title: Increasing the Use of Donated Embryos: A Demonstration
Brief Title: Frozen Embryo Donation Study
Acronym: FREDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston IVF (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Brandeis University (Other)
Responsible Party: Principal Investigator, Alison Zimon, Reproductive Endocrinologist, Boston IVF
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FREDS; EAAPA111016 (Other Grant/Funding Number: Department of Health and Human Services)
Record Dates: First submitted 2013-05-21; First posted 2013-06-21 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: In Vitro Fertilization (IVF); Embryo donation
MeSH Terms: conditions — Infertility | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced clinic-based support/counseling (Experimental): Scheduling a consult with a licensed social worker to discuss embryo disposition options. Additional enhanced support services and educational services provided by embryologists, nurses and physicians in the Frozen Embryo Donation Service will be offered.
  Interventions: Other: Enhanced clinic-based support/counseling
- Patients receiving standard of care (Active Comparator): Patients who receive standard of care regarding embryo disposition options
  Interventions: Other: Control

INTERVENTIONS:
Other: Enhanced clinic-based support/counseling — Additional enhanced support services and educational services provided by embryologists, nurses and physicians in the Frozen Embryo Donation Service will be offered.
  Arms: Enhanced clinic-based support/counseling
Other: Control
  Arms: Patients receiving standard of care

SUMMARY:
The purpose of this study is to improve patient understanding of and interest in donating frozen embryos resulting from in vitro fertilization (IVF) to others undergoing infertility treatment.

DETAILED DESCRIPTION:
The first phase of this study involves the mailing of a survey to current Boston IVF patients who have embryos frozen in storage. A survey will be sent to these individuals to assess their knowledge and understanding of frozen embryos and if they would be interested in embryo donation.

The second phase of research will randomize these patients into two groups: control and intervention. The control groups will receive their standard of treatment regarding frozen embryos, which consists of receiving a yearly storage bill. The intervention group will receive a letter from their physician of record and a follow up phone call from a research assistant offering the opportunity to schedule a consult with a licensed social worker at Boston IVF. The consult is meant to serve as a chance to discuss the difficult decision around embryo disposition. The consult for these patient will be free of charge, covered with funds from our grant. Additional enhanced support services and educational services provided by embryologists, nurses and physicians in the Frozen Embryo Donation Service will be offered. These enhanced services will also be free of charge to subjects.

The third phase of the study includes the mailing of a letter to a random sample of patients with embryos frozen in storage at Boston IVF. This letter will be an invitation to contact Boston IVF to schedule a consult with a licensed social worker to discuss embryo disposition options. The consult for these patient will be free of charge, covered with funds from our grant.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Boston IVF with embryos frozen in storage

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3568 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Increase in embryo donation | Approximately 2 years
  We will be tracking to see if there is an increase in embryo donation as a result of the study

CONTACTS AND LOCATIONS:
Overall Officials: Alison Zimon, MD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

REFERENCES:
- [Derived] Zimon AE, Shepard DS, Prottas J, Rooney KL, Ungerleider J, Halasa-Rappel YA, Sakkas D, Oskowitz SP. Embryo donation: Survey of in-vitro fertilization (IVF) patients and randomized trial of complimentary counseling. PLoS One. 2019 Aug 15;14(8):e0221149. doi: 10.1371/journal.pone.0221149. eCollection 2019. PMID 31415660